CLINICAL TRIAL: NCT05274087
Title: A Randomized, Double-Blind, Three-Period Crossover Study to Evaluate the Effect of Different Warm-Up Times of Risankizumab Autoinjector (AI) on the Injection Pain Experiences in Healthy Volunteers
Brief Title: Study to Evaluate the Effect of Different Warm-Up Times of Risankizumab Autoinjector (AI) on the Injection Pain Experiences in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M20-200
Record Dates: First submitted 2022-03-08; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Risankizumab
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (Experimental): Participants will receive Regimen A (15-minute autoinjector (AI) warm-up time) in Period 1, Regimen B (30-minute AI warm-up time) in Period 2 followed by Regimen C (45-minute AI warm-up time) in Period 3.
  Interventions: Drug: Risankizumab
- Group 2 (Experimental): Participants will receive Regimen B in Period 1, Regimen C in Period 2 followed by Regimen A in Period 3.
  Interventions: Drug: Risankizumab
- Group 3 (Experimental): Participants will receive Regimen C in Period 1, Regimen A in Period 2 followed by Regimen B in Period 3.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous autoinjector
  Other Names: SKYRIZI

SUMMARY:
The objective of this study is to assess the impact of different warm-up times of risankizumab autoinjector (AI) on the participant injection site pain experience in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index (BMI) is >= 18.0 to <= 30.0 kg/m2.

Exclusion Criteria:

* Any findings in the medical examination that are deviating from normal and judged as clinically relevant by the investigator.
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease judged as clinically relevant by the investigator.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, or psychiatric disease or disorder, or any other uncontrolled medical illness.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Change in Injection Site Pain Assessed Using Visual Analog Scale | Up to approximately 15 days
  Injection site-related pain assessments will be recorded directly by the participant using a VAS after the injection is complete (within approximately 5 minutes and 1 hour post-dose).
Percentage of Participants Experiencing Adverse Events | Up to approximately 155 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

SECONDARY OUTCOMES:
Participant Rated Acceptability Assessed as Change in Self-Injection Assessment Questionnaire (SIAQ) | Up to approximately 15 days
  SIAQ is an electronic patient-reported outcomes (ePRO) device assessing participant acceptability with scores ranging from 0 (worst experience) to 10 (best experience).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 223662, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No